CLINICAL TRIAL: NCT06460220
Title: SAFETY-Parent: Online Learning Module to Support Parents of Suicidal Youth
Acronym: SAFETY-P
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Hughes (Other)
Collaborators: American Foundation for Suicide Prevention (Other)
Responsible Party: Sponsor-Investigator, Jennifer Hughes, Psychologist & Clinical Scholar, Associate Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003043
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Suicide; Suicide, Attempted; Suicide and Self-harm; Suicide Threat
MeSH Terms: conditions — Suicide; Suicide, Attempted; Self-Injurious Behavior | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Phase 2 will include pilot testing of the SAFETY-P asynchronous parent intervention module with a nonrandomized case series of 10 families receiving services in CATC.
  Phase 3 will include an RCT with N = 30 youth and parents, who will be randomized either to SAFETY-P + treatment as usual (TAU) or to TAU alone.
Who Masked: Outcomes Assessor
Masking Description: Independent evaluators, masked to condition, will conduct outcome assessments with parents and youth at baseline,1-month (the typical length of TAU in CATC prior to linking youth patients to ongoing outpatient care), and 3-month follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safe Alternatives for Teens and Youth - Parent (SAFETY-P) + Treatment as Usual (TAU) (Experimental): Phase 2 will include pilot testing of the SAFETY-P asynchronous parent intervention module with a nonrandomized case series of 10 families receiving services in CATC. Participants will be provided with the SAFETY-P modules and complete follow-up measures after one month.
  Phase 3 will include an RCT with N = 30 youth and parents, with half randomized to SAFETY-P + treatment as usual (TAU). Participants will complete measures at baseline, 1 month, and 3 months.
  Interventions: Behavioral: Safe Alternatives for Teens and Youth - Parent (SAFETY-P); Behavioral: Treatment As Usual (TAU)
- Treatment As Usual (TAU) (Other): Phase 3 will include an RCT with N = 30 youth and parents, with half randomized treatment as usual (TAU). Participants will complete measures at baseline, 1 month, and 3 months.
  Interventions: Behavioral: Treatment As Usual (TAU)

INTERVENTIONS:
Behavioral: Safe Alternatives for Teens and Youth - Parent (SAFETY-P) — The parent component of SAFETY focuses on enhancing parents' skills in supporting youth safety and managing parental distress during a suicidal crisis, ideal content to adapt for web-based delivery for parents. Specifically, parent information includes psychoeducation about suicide risk and protective factors, lethal means restriction, development of a parent distress tolerance plan (i.e., Parent Safety Plan), parent self-care and sources of support, strengthening the youth/parent relationship, and focus on care linkage for the youth. The SAFETY-P asynchronous parent intervention module will include text, interactive handouts, vignettes, and short video examples. The SAFETY-P module will allow for parents to access information and skills training on their own time, with the opportunity and encouragement to ask informed questions of their child's clinician; this will provide clinicians the opportunity to utilize their check-ins with parents more effectively to address youth safety.
  Arms: Safe Alternatives for Teens and Youth - Parent (SAFETY-P) + Treatment as Usual (TAU)
Behavioral: Treatment As Usual (TAU) — TAU will consist of treatment and case management as usual in the NCH Critical Assessment and Treatment (CATC) program. This may include individual and group therapy sessions for the youth, family therapy, medication management, and case management/discharge planning. Frequency of these services varies by availability and care linkage to ongoing outpatient care. We will track the number, type and length of all treatment and case management services provided as part of TAU in CATC to control for time spent in by parents and youth in TAU across study conditions. Additionally, the Child and Adolescent Services Assessment (CASA), a services use measure, will be utilized to capture any additional treatments and parents' involvement in those treatments.

SUMMARY:
This project aims to adapt the parent component of Safe Alternatives for Teens and Youth (SAFETY) outpatient intervention to SAFETY-Parent (SAFETY-P), a self-paced interactive learning module for parents, to be implemented as an augmentation for youth being seen for suicidal ideation, suicidal behavior, or recent suicide attempts across multiple settings at Nationwide Children's Hospital (NCH, Columbus, Ohio).

DETAILED DESCRIPTION:
This research project has iterative aims focused on the development and pilot testing of the SAFETY-P asynchronous parent intervention module. Phase 1 will focus on finalizing SAFETY-P content for the online learning module. Phase 2 will be a small open case series integrating additional key stakeholder feedback via formative usability testing. Phase 3 will test the revised module in a pilot RCT, to establish methods and protocols for a future large-scale clinical trial.

Phase 1/Aim 1 (Intervention Adaptation for Online Delivery): Phase 1 will include 4 separate stakeholder focus groups (adolescents, parents, behavioral health [BH] inpatient and outpatient providers, and parent survivors of suicide loss) to advise on adaptations to SAFETY-P and development of the self-paced, interactive module to be used in Phase 2.

Aim 1: Adapt the parent component of SAFETY to content for the SAFETY-P asynchronous parent intervention module and determine feasibility and acceptability of SAFETY-P to this asynchronous module delivery.

Hypothesis (Hyp) 1.1: SAFETY content will be adapted successfully to SAFETY-P; stakeholders will report that use of an online asynchronous learning module for parents is feasible and acceptable based on qualitative coding outcomes.

Phase 2/Aim 1 (Case Series Iterative Adaptation): Phase 2 will include pilot testing of SAFETY-P with a nonrandomized case series of 5 clinicians and 10 families. Participants will be invited to use SAFETY-P for up to one month. Feedback from this case series will inform iterative adaptations to the SAFETY-P module.

Hyp 1.2: SAFETY-P will be feasible to use (parents will report using SAFETY-P at least twice during the one month, clinicians will report discussing SAFETY-P content with parents at least once during the one month).

Hyp 1.3: Parents and clinicians will report that use of SAFETY-P is acceptable via formative usability testing interview feedback and on measures of acceptability (System Usability Questionnaire rating of >68; Mobile Application Rating Scale: User Version (uMARS) acceptable scores ≥ 3).

Phase 3/Aims 2-4 (Pilot RCT of SAFETY-P): To assess feasibility and acceptability of SAFETY-P, we will conduct a pilot RCT with N=30 youth and parents, who will be randomized to either SAFETY-P + treatment as usual (TAU) or to TAU alone.

Aim 2: Conduct a pilot study of SAFETY-P. Outcomes will include study recruitment and retention rates, SAFETY-P parent satisfaction ratings, clinician-report of SAFETY-P use and effectiveness, and adverse event reports.

Hyp 2.1: The sample can be recruited in 1 year. Hyp 2.2: >80% will participate throughout the 3 months. Hyp 2.3: Parents will report using SAFETY-P ≥ 2 times. Hyp 2.4: Parents will report high satisfaction on the SAFETY-P Satisfaction Scale (acceptable item scores ≥ 3) and the Peabody Treatment Progress Battery, Service Satisfaction Scale (acceptable item scores ≥ 3).

Hyp 2.5: Clinicians will report high satisfaction on the SAFETY-P Satisfaction Scale (acceptable item scores ≥ 3).

Exploratory Aim 3 (Parent Outcomes): Investigate if SAFETY-P leads to changes parent functioning (the intervention "target") - at 1 and 3-month follow-up, we will measure between-group differences.

Hyp 3.1: SAFETY-P+TAU parents will have preferential outcomes on: a) parent emotion regulation, b) parent depressive symptoms, c) caregiver strain, d) family conflict, e) parent perceived self-efficacy to manage their child's suicidal crises, and f) parent expectations of adolescents' risk.

Exploratory Aim 4 (Youth Outcomes): Explore preliminary effectiveness of the SAFETY-P at decreasing youth suicide risk factors - we will measure between-group differences at 1 and 3-month follow-up.

Hyp 4.1: SAFETY-P+TAU youth will have preferential outcomes on: a) youth suicidal ideation (SI), b) suicide attempts (SA), c) non-suicidal self-injury (NSSI), d) and services use (including TAU sessions attended and use of higher levels of care for suicidal crises such as emergency department or inpatient hospitalization), e) family conflict, f) thwarted belongingness, and g) perceived burdensomeness.

ELIGIBILITY:
Inclusion Criteria:

For Phase 1 interviews and focus groups:

1. Youth or young adults (<25 years) with prior suicidal ideation or suicide attempts; parents whose child had a history of suicidal ideation and/or suicide attempt before age 18; medical or behavioral health provider of suicidal youth; and parents whose child died from suicide before age 18

For Phase 2 and the Phase 3:

1. Youth is currently in treatment with the Critical Assessment and Treatment Clinic (CATC) at NCH for suicidal thoughts or behaviors
2. Youth is between the ages of 10-18 (18-year-old youth must still be in high school and living at home with parents for duration of the study)
3. At least one parent is able to participate
4. Youth and parent are fluent in English

Exclusion Criteria:

For all four Phase 1 groups:

1. Cannot read or speak English (given focus group to be conducted in English

For Phase 2 and Phase 3 participants:

1. The youth or parent has an acute psychiatric or medical condition that would interfere with their ability to participate in study procedures
2. Lack of access to a digital device (smartphone, iPad, tablet computer, desktop, laptop PC)

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with intervention on the Peabody Treatment Progress Battery (PTPB) - Service Satisfaction Scale (SSS) | 1 month, 3 months
  The PTPB is an integrated set of brief, reliable, and valid instruments that can be administered efficiently at low cost and can provide systematic feedback for use in treatment planning. It includes eleven measures completed by youth, caregivers, and/or clinicians that assess clinically-relevant constructs such as symptom severity, therapeutic alliance, life satisfaction, motivation for treatment, hope, treatment expectations, caregiver strain, and service satisfaction. The SSS provides a general indicator of how well youth and adult caregivers perceive the mental health organization's services.
Use of intervention as measured by information provided by the Brainer Learning Management System (LMS) | 1 month, 3 months
  The LMS provides data on which components of the SAFETY-P modules were accessed, completion or non-completion of the component module, at which point in the content does discontinuation occur, time spent using the modules.
Intervention feasibility and acceptability on the SAFETY-P Satisfaction Scale | 1 month, 3 months
  The SAFETY-P Satisfaction Scale consists of 8 items and measures acceptability of the SAFETY-P tool.
Intervention usability on the System Usability Scale | 1 month
  The System Usability Scale consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. The scale evaluates a wide variety of products and services, including hardware, software, mobile devices, websites and applications.
Intervention acceptability on the Mobile Application Rating Scale: User Version (uMARS) | 1 Month
  The uMARS is a simple tool that can be reliably used by end-users to assess the quality of mHealth apps. The uMARS provides a 20-item measure that includes 4 objective quality subscales-engagement, functionality, aesthetics, and information quality-and 1 subjective quality subscale.
Utilization of mental health services on the Child and Adolescent Services Assessment: Brief and Adapted version (CASA) | Baseline, 1 month, 3 months
  The CASA is a self and parent report instrument designed to assess the use of mental health services by children aged 8-18 yrs. The CASA includes 31 settings covering inpatient, outpatient, and informal services provided by a variety of child serving providers and sectors. It collects information on whether a service was ever used and more detailed information (length of stay/number of visits, focus of treatment) on services used in the recent past.

SECONDARY OUTCOMES:
Change from baseline in suicidal ideation and behavior on the Columbia-Suicide Severity Rating Scale (C-SSRS) at 30 days and 3 months | Baseline, 1 month, 3 months
  The C-SSRS is a validated, semi-structured interview that assesses both suicidal behavior and suicidal ideation (yes/no, frequency), with flexible time points and multiple informants depending on administrator purpose and need.
Change from baseline in suicidal ideation severity on the Suicidal Ideation Questionnaire-Junior (SIQ-JR) at 1 month and 3 months | Baseline, 1 month, 3 months
  The SIQ-JR is a 15-item modified version of the 30-item Suicidal Ideation Questionnaire. The SIQ-JR is a validated self-report measure of suicidal ideation severity in adolescents (7-point scale; 0="I never had this thought"; 6="Almost every day").
Youth psychopathology as measured by the Child Behavior Checklist (CBCL) | Baseline
  The CBCL is a standardized measure based on new national norms that were collected February 1999-January 2000. The CBCL is to be completed by the parent/caretaker who spends the most time with the child. The CBCL provides ratings for 20 competence and 120 problem items. The CBCL includes open-ended items covering physical problems, concerns, and strengths. Parents rate how true each item is now, or was within the past 6 months. The CBCL yields scores on internalizing, externalizing, and total problems as well as scores on DSM-IV related scales.
Youth psychopathology as measured by the Youth Self-Report (YSR) | Baseline
  The Youth Self-Report (YSR) is a widely used child-report measure that assesses problem behaviors along two "broadband scales": Internalizing and Externalizing. It also scores eight empirically based syndromes and DSM-oriented scales, and provides a summary of Total Problems. The measure assesses "Total Competency," which is a scale comprised of competency in activities, social functioning, and school performance.
Change from baseline in depressive symptoms for youth and parent participants on the Center for Epidemiological Studies Depression Scale (CES-D) at 1 month and 3 months | Baseline, 1 month, 3 months
  The CES-D is a 20-item measure that asks caregivers to rate how often over the past week they experienced symptoms associated with depression, such as restless sleep, poor appetite, and feeling lonely. Response options range from 0 to 3 for each item (0 = Rarely or None of the Time, 1 = Some or Little of the Time, 2 = Moderately or Much of the time, 3 = Most or Almost All the Time). Scores range from 0 to 60, with high scores indicating greater depressive symptoms.
Change from baseline in feelings of which measures thwarted belongingness and perceived burdensomeness for youth participants on the Interpersonal Needs Questionnaire-Adolescent Version (INQ) at 1 month and 3 months | Baseline, 1 month, 3 months
  The INQ-15 (19) is a self-report measure composed of 15 items that evaluate the main constructs of interpersonal suicide theory (8): perceived burdensomeness and thwarted belongingness. The items are answered on a 1-7 Likert scale (1 = Not at all true for me, 4 = Somewhat true for me, 7 = Very true for me).
Change from baseline in parent emotional dysregulation on the Difficulties in Emotion Regulation Scale (DERS) at 1 month and 3 months | Baseline, 1 month, 3 months
  The DERS is a brief, 36-item, self-report questionnaire designed to assess multiple aspects of emotion dysregulation. The measure yields a total score as well as scores on six scales derived through factor analysis.
Parent psychopathology as measured by the Brief Symptom Inventory (BSI) | Baseline
  The BSI is a 53-item self-report inventory in which participants rate the extent to which they have been bothered (0 ="not at all" to 4="extremely") in the past week by various symptoms. The BSI has nine subscales designed to assess individual symptom groups: somatization, obsessive-compulsive, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, and psychoticism. The BSI also includes three scales that capture global psychological distress.
Change from baseline in parent distress related to caring for a child with mental illness on the Caregiver Strain Questionnaire at 1 month and 3 months | Baseline, 1 month, 3 months
  The Caregiver Strain Questionnaire is a 21-item measure of self-reported strain experienced by caregivers and families of youth with emotional problems, with responses on a 5-point Likert scale (0 = Not at all, 4 = very much). It assesses the demands, responsibilities, difficulties, and negative psychological consequences of caring for children and adolescents with emotional and behavioral disorders.
Change from baseline in parental confidence in their ability to prevent or manage a suicidal crisis on the Parent Self-Efficacy for Suicide and the Self-Assessed Expectations of Suicide Risk Scale, Adapted for Parents at 1 month and 3 months | Baseline, 1 month, 3 months
  The Parent Self-Efficacy for Suicide and the Self-Assessed Expectations of Suicide Risk Scale is a 12 item measure using a 10-point Likert scale (0=not at all confident, 5=somewhat confident, 10=completely confident). It measures parental confidence in caring for an adolescent experiencing suicidal ideation.
Change from baseline in family conflict measures on the Conflict Behavior Questionnaire (CBQ) at 1 month and 3 months | Baseline, 1 month, 3 months
  The Conflict Behavior Questionnaire (CBQ) is designed to obtain evaluations of parent and adolescent behavior directly from parent and adolescent. The questionnaire reliably measures whether or not a family is experiencing distress.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer L Hughes, PhD, MPH, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No